CLINICAL TRIAL: NCT05224011
Title: A Prospective Study to Evaluate the Safety and Effectiveness of the Boppli™ in Measuring Mean Arterial Pressure (MAP), Systolic Blood Pressure (SBP), and Diastolic Blood Pressure (DBP) as Compared to an Invasive Arterial Reference
Brief Title: Non-invasive Continuous Blood Pressure Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PyrAmes Inc. (Industry)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PyrAmes-2021-01
Record Dates: First submitted 2022-01-04; First posted 2022-02-04 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-06

CONDITIONS: Blood Pressure
Keywords: Neonates; Blood Pressure monitoring; Medical Device; Non-Invasive Blood Pressure Monitoring; Invasive Arterial Lines

STUDY DESIGN:
Intervention Model Description: The study is a single-arm study in which patient measurements will be obtained using both the investigational device-Boppli-as well as traditional blood pressure measurement collected via IAL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): The Boppli device will be applied to the patients' arm or foot on either side of the body and is intended for single use of up to 72 hours and is discarded following use. The device will only be used in patients requiring continuous blood pressure monitoring, through the use of an invasive arterial line (IAL), to compare the data obtained by the Boppli to that obtained by the IAL.
  Interventions: Device: Boppli Infant Blood Pressure Monitor

INTERVENTIONS:
Device: Boppli Infant Blood Pressure Monitor — The intervention is a medical device for the non-invasive measurement of blood pressure in infants

SUMMARY:
The Boppli device was designed to provide continuous non-invasive blood pressure (cNIBP) monitoring for infants, including neonates, in intensive care settings by detecting systolic, diastolic, and mean arterial blood pressure values comparable to that of an invasive arterial line (IAL) within published accuracy criteria. The device consists of an array of capacitive sensors contained in a soft, flexible, biocompatible band. It applies proprietary algorithms to capacitance detections to generate accurate systolic, diastolic, and mean arterial blood pressure and waveform data, then communicates the data to an external device via Bluetooth Low Energy for storage and display. It may be applied to the patient's arm or foot on either side of the body, which is advantageous for infants whose bodies provide limited surface area for medical devices or equipment. It does not require high skin pressure when correctly placed. The device is intended for single use of up to 72 hours and is discarded following use.

DETAILED DESCRIPTION:
The purpose of this study is to validate PyrAmes's non-invasive blood pressure measurements against invasive blood pressure measurements taken with a reference device that is routinely used in a hospital setting, is generally regarded as accurate, and is routinely used in the diagnosis and treatment of patients. In this case, the reference device is the invasive arterial line, which is routinely used in the care of infants in intensive care settings to collect accurate, continuous invasive blood pressure measurements.

The specific aim of this study is to record data obtained by use of the Boppli device, along with invasive measurements of blood pressure, for use in validating the Boppli device measurements and algorithm. The changes in capacitance will serve as an input for the Boppli algorithm and systolic, diastolic, and mean arterial pressure will be output. The measurements generated from the non-invasive Boppli Device will be validated against the invasive measurements from the reference device. This is a prospective, multi-center clinical study to validate the effectiveness of the Boppli Blood Pressure Monitor as compared to an invasive arterial reference. The study will evaluate the accuracy and precision of the Boppli system for continuous blood pressure monitoring by comparing SBP (systolic blood pressure), DBP (diastolic blood pressure), and MAP (mean arterial pressure) against the reference methodology.

Invasive arterial lines (IAL) were selected as the comparator for this study. IALs are the current gold standard for continuous blood pressure monitoring for infants in intensive care settings. Sphygmomanometers are widely used for non-invasive blood pressure monitoring among other populations but have documented issues with accuracy in patients with very low blood pressures, which includes many neonates and pediatric patients. Due to their potentially low accuracy in detecting blood pressure in infants, the manual sphygmomanometer is not regarded as an appropriate comparator for the Boppli device.

As stated in reference standards ISO 81060-2 and ANSI SP10, intra-arterial methods should not be used for subjects solely for the purpose of validating instrument performance. However, the SP10 standard states that in validation studies in children less than 3 years of age, the intra-arterial method should be used as the reference standard. In addition, it is noted that ISO 81060-2 explicitly states that children less than 3 years of age should not be included in clinical investigations using auscultatory reference readings. Therefore, this study will be conducted on clinical subjects (neonates/infants) in whom an intra-arterial line has already been placed for reasons other than validating instrument performance.

Primary objective: To assess the accuracy and precision of the Boppli system in measuring SBP, DBP, and MAP as compared to an invasive arterial line for continuous blood pressure monitoring.

Secondary Objective: To assess the safety of the Boppli system in a clinical setting.

Methods: Data to assess device efficacy, subject safety, and subject demographics will be collected from the Investigational sites. Data will be collected using an electronic data collection system (EDC) designed to comply with 21 CFR Part 11 and will be recorded into the electronic Case Report Form (eCRF). Primary source documentation will come directly from the subject's medical record

ELIGIBILITY:
Inclusion Criteria:

Groups 1 - 4:

* Pediatric patients less than 1 year of age and less than 5000 g in weight (primary target)
* Requires intra-arterial blood pressure monitoring

Group 5:

* Pediatric patients
* Requires intra-arterial blood pressure monitoring

NOTE: Under no circumstance should an invasive arterial line be implanted in a patient due to this study, if not medically necessary.

Exclusion Criteria:

* Skin conditions that limit the placement of the device
* Patients connected to or treated by other devices that may alter the pulse waveform
* Patients with a cardiac or vascular malformation that results in an abnormal waveform inappropriate to be considered a reference standard.

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Assess the accuracy and precision of the Boppli System in continuous blood pressure monitoring | 6 - 72 Hours
  The primary objective of this pivotal study is to assess the accuracy and precision of the Boppli system in measuring systolic blood pressure (SBP), diastolic blood pressure (DBP) and mean arterial pressure (MAP), as compared to an invasive arterial line for continuous blood pressure monitoring in infants.
  The following steps will be performed specifically to collect data for this study:
  * Boppli will be used alongside IALs onsite to collect blood pressure measurements, as well as pulse waveforms.
  * Continuous data from the IAL and Boppli will be paired for comparison
  * The total duration of data collection is expected to be approximately 6 hours with some patients remaining in the study up to 72 hours. However, subjects will not be required to remain in the study should clinical care indicate that the IAL should be removed.
  * Observed rapid changes in blood pressure will be collected and the Boppli's accuracy in detecting these changes will be compared against IAL

SECONDARY OUTCOMES:
Assess the safety of the Boppli System in a clinical setting | 6 - 72 Hours
  The secondary objective is to assess the safety of the Boppli System in a clinical setting. This will be done by collecting and analyzing all adverse events observed during the study. Information on the usability of the device and its impact on workflow will also be collected.
  The following steps will be performed specifically to collect data for this study:
  * Boppli will be used alongside IALs onsite to collect blood pressure measurements, as well as pulse waveforms.
  * Continuous data from the IAL and Boppli will be paired for comparison
  * The total duration of data collection is expected to be approximately 6 hours with some patients remaining in the study up to 72 hours. However, subjects will not be required to remain in the study should clinical care indicate that the IAL should be removed.
  * Observed rapid changes in blood pressure will be collected and the Boppli's accuracy in detecting these changes will be compared against IAL

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Yusuf, Ph.D., Principal Investigator — University of Calgary - Department of Pediatrics
Locations (1):
- Foothills Medical Center Neonatal Intensive Care Unit, NICU 51, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No